CLINICAL TRIAL: NCT00113646
Title: Non-Myeloablative HLA-Mismatched Ex-Vivo T-cell Depleted Stem Cell Transplantation for Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Expiration of MEDI-507
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Thomas Spitzer, Director Cellular Therapy and Transplantation Laboratory, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-163
Record Dates: First submitted 2005-06-09; First posted 2005-06-10 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Lymphoma; Leukemia; Multiple Myeloma; Myelodysplastic Syndrome
Keywords: Non-Myeloablative; T-cell Depleted; Mismatched; Stem Cell Transplantation
MeSH Terms: conditions — Lymphoma; Leukemia; Multiple Myeloma; Myelodysplastic Syndromes | interventions — siplizumab

INTERVENTIONS:
Drug: MEDI-507 — MEDI-507 0.1 mg/kg on transplant day-8, 0.6 mg/kg on days-7 and -6
Procedure: Non-myeloablative Ex-Vivo T-cell Depleted PBSC Transplant — Cyclophosphamide 60 mg/kg on transplant days -7 and -6; Fludarabine 25 mg/m2 days -5,-4,-3,-2,-1; MEDI-507 0.1 mg/kg on day -8, 0.6 mg/kg on days -7,-6

SUMMARY:
The purpose of this study is to determine if recipients of non-myeloablative ex-vivo T-cell depleted peripheral blood (PBSC) stem cell transplantation using a mismatched related donor will have less severe graft versus host disease (GVHD), transplant related mortality, and less graft failure compared to alternative haploidentical stem cell transplantation.

DETAILED DESCRIPTION:
One major obstacle to further advancement in the role of bone marrow transplant (BMT) in hematological malignancies is graft-versus-host-disease (GVHD), which can best be prevented by removing T-cells from the donor stem cell product. However, previous experience with T-cell depletion has been associated with an increased rate of engraftment failure and leukemic relapse. Another obstacle is that a large fraction of leukemia and lymphomas afflict older patients who are more prone to GVHD and have co-morbid conditions that prevent them from being a candidate for BMT.

This trial uses a non-myeloablative conditioning regimen with cyclophosphamide, MEDI-507, fludarabine, and thymic irradiation followed by a T-cell depleted PBSC infusion. Cyclosporine is used for GVHD prophylaxis, and tapered beginning on day 35. Data from our mouse model and previous clinical trials have demonstrated that this approach can induce mixed chimerism without GVHD, with the potential for conversion of mixed chimerism to full donor hematopoiesis following donor leukocyte infusions.

ELIGIBILITY:
Inclusion Criteria:

* Disease Status: NHL, HD, MM that are chemorefractory or relapsed; CLL that is Rai stage III or IV, or lymphocyte doubling time of 6 months, or stage I/II resistant to > 2 cycles of chemotherapy regimens; CML in accelerated or blast phase; MDS with life-threatening cytopenias; patients who have had a previous autologous or allogeneic bone marrow or stem cell transplant; other hematological disorders where allogeneic transplant is appropriate and the risk of conventional transplantation is considered to be unacceptably high.
* estimated disease free survival of less than one year
* ECOG performance status of 0, 1, or 2
* HLA 1 to 3 mismatched (at A, B, DR loci) related donor

Exclusion Criteria:

* Cardiac disease: symptomatic congestive heart failure, ejection fraction of < 45%, active angina pectoris or uncontrolled hypertension.
* Pulmonary disease: severe chronic obstructive lung disease, or symptomatic restrictive lung disease, or corrected DLCO of < 50%
* Renal disease: serum creatinine > 2.0 mg/dl or creatinine clearance < 50 ml/min
* Hepatic disease: serum bilirubin > 2.0 mg/dl or alkaline phosphate, SGPT or SGOT > 3 x normal
* Neurologic disease: symptomatic leukoencephalopathy, active CNS malignancy or other neuropsychiatric abnormalities believed to preclude transplantation
* HIV antibody or Hepatitis B surface antigen positivity
* Uncontrolled infection
* Presence of HAMA or HAHA in patient previously treated with monoclonal antibody therapy or who have received a product in which the preparation involved a monoclonal antibody affinity step

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2002-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the risk of graft loss and severe GVHD or transplant related mortality at < 100 days following HLA-mismatched non-myeloablative stem cell transplantation. | 36 months

SECONDARY OUTCOMES:
To evaluate progression free and overall survival following HLA mismatched non-myeloablative stem cell transplantation for hematologic malignancy. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Spitzer, M.D., Principal Investigator — Massachusetts General Hospital, Harvard University
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States